CLINICAL TRIAL: NCT05762107
Title: A Phase 2a Randomized, Double-blind, Placebo-controlled, Multiple-dose, Crossover Study of the Effect of ZT-01 on Frequency of Nocturnal Hypoglycemia in Type 1 Diabetes Mellitus
Brief Title: A Study of the Effect of ZT-01 on Night-time Hypoglycemia in Type 1 Diabetes
Acronym: ZONE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zucara Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ZT01-CL-2001
Record Dates: First submitted 2023-02-27; First posted 2023-03-09 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Type 1 Diabetes Mellitus With Hypoglycemia
Keywords: nocturnal hypoglycemia

STUDY DESIGN:
Intervention Model Description: The participant will be randomized to receive placebo and one of three dose levels of ZT-01 in a crossover design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ZT-01 7 mg (Experimental): Participants receive placebo and ZT-01 7 mg each by subcutaneous injection daily for 28 days, randomized to order
  Interventions: Drug: Placebo; Drug: ZT-01, 7 mg
- ZT-01 15 mg (Experimental): Participants receive placebo and ZT-01 15 mg by subcutaneous injection daily for 28 days, randomized to order
  Interventions: Drug: Placebo; Drug: ZT-01, 15 mg
- ZT-01 22 mg (Experimental): Participants receive placebo and ZT-01 22 mg by subcutaneous injection daily for 28 days, randomized to order
  Interventions: Drug: Placebo; Drug: ZT-01, 22 mg

INTERVENTIONS:
Drug: Placebo — Subject receives Placebo by subcutaneous injection daily for 28 days
Drug: ZT-01, 7 mg — Subject receives ZT-01 7 mg by subcutaneous injection daily for 28 days
  Arms: ZT-01 7 mg
Drug: ZT-01, 15 mg — Subject receives ZT-01 15 mg by subcutaneous injection daily for 28 days
  Arms: ZT-01 15 mg
Drug: ZT-01, 22 mg — Subject receives ZT-01 22 mg by subcutaneous injection daily for 28 days
  Arms: ZT-01 22 mg

SUMMARY:
The goal of this clinical trial is to learn about the effect of the study drug (ZT-01) on low blood sugar (hypoglycemia) in adults with type 1 diabetes (T1D) who have been having low blood sugars ("hypos") at night. ZT-01 increases the amount of a hormone called glucagon during low blood sugar, and this may help prevent the occurrence of hypos. The main questions this trial aims to answer are whether ZT-01 lowers the number of hypos happening at night, and what its effects are on blood sugar levels. The safety of ZT-01 will also be measured.

Participants will be asked to wear a study-provided continuous glucose monitor (CGM) during two 4-week periods when they will self-inject the study drug before bed. They will get ZT-01 at one of three dose levels during one period, and placebo (which looks like the study drug but doesn't contain the active ingredient) during the other. Neither the participant nor the study site will know what they are receiving during each treatment period or see data from the CGM. The participant will continue to use their usual methods of measuring blood sugar (including their personal CGM) and giving insulin during the study. The participant will be asked to complete a short diary each evening, and will be asked to upload the CGM data to a study phone every day.

If a participant uses their own CGM and is willing to share information on how often they have low blood sugar with the study site at the first visit to see if they meet study entry requirements, they will have 6 study visits, 2 study phone calls, and be in the study for about 16 weeks. If they don't use CGM or don't want to share their information, then they will be asked to wear a study CGM for an extra 4 weeks to find out how many low blood sugars they have, and will have an extra visit.

Study participants will be asked to give blood and urine for testing to see whether they meet the requirements to enter the study, and at the start and end of each treatment period to see if the study treatment has any effects. They will also have their blood pressure and temperature taken at each study visit, and have an ECG at 4 visits to measure the electrical activity of their heart.

Some participants will be asked to also take part in a sub-study where their blood level of ZT-01 and glucagon is measured, after the first and last dose. They will be asked to stay at the study site overnight for each set of measurements (4 in total).

ELIGIBILITY:
Inclusion Criteria:

* Has type 1 diabetes for at least 5 years
* is at risk of nocturnal hypoglycemia (if using personal CGM, time below 54 mg/dL at least 1% over previous 4 weeks at screening; if not using personal CGM then recent history suggestive of nocturnal hypoglycemia at screening and time below 54 mg/dL at least 1% over 4 weeks using blinded study CGM during additional screening)
* HbA1c at screening </= 10.0%
* Body mass index (BMI) at screening >/=18.5 to <33 kg/m2

Exclusion Criteria:

* Has been hospitalized for diabetic ketoacidosis (DKA) more than once within previous 6 months
* Has experienced >/= 1 severe hypoglycemia (requiring assistance) during previous 4 weeks or >2 in previous 3 months
* Diagnosis of type 2 diabetes, pheochromocytoma, insulinoma, glucagonoma, acromegaly, Cushing's disease, glycogen storage disease, adrenal insufficiency
* Clinically significant kidney disease
* Abnormal liver function

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2023-07-28 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of nocturnal hypoglycemia | During each 28 day treatment period
  Rate of nocturnal (midnight to 06:00 AM) hypoglycemic events (glucose <54 mg/dL) lasting at least 15 minutes, compared to placebo

SECONDARY OUTCOMES:
Incidence and severity of adverse events (AEs) | During each 28 day treatment period and 2-week followup
  Number of patients experiencing AEs compared to placebo
Glucose time below range | During each 28 day treatment period
  Glucose time below 54 mg/dL (as %) compared to placebo
Incidence of hypoglycemia | During each 28 day treatment period
  Number of hypoglycemic events (glucose <70 mg/dL for at least 15 minutes, compared to placebo

OTHER OUTCOMES:
Glucose time in range | During each 28-day treatment period
  Glucose time in range (70-180 mg/dL, %) compared to placebo
Mean glycemic variability | During each 28 day treatment period
  Percent coefficient of variation of glucose values compared to placebo
Mean glucose concentration | During each 28 day treatment period
  Mean glucose concentration compared to placebo

CONTACTS AND LOCATIONS:
Locations (33):
- United States (26):
  - Headlands Research, Escondido, California
  - USC Keck Medicine Eastside Center for Diabetes, Los Angeles, California
  - LCGK Research, San Carlos, California
  - East Coast Institute for Research LLC, Jacksonville, Florida
  - Suncoast Clinical Research, New Port Richey, Florida
  - Hanson Diabetes Center, Port Charlotte, Florida
  - Metabolic Research Institute, West Palm Beach, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Physicians Research Associates LLC, Lawrenceville, Georgia
  - East Coast Institute for Research, Macon, Georgia
  - IU Health University Hospital, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Baltimore VA Medical Center, Baltimore, Maryland
  - MedStar Good Samaritan Hospital, Baltimore, Maryland
  - Elite Research Center, Flint, Michigan
  - Palm Research Center, Inc., Las Vegas, Nevada
  - Albany Medical Center, Albany, New York
  - NYC Research Inc., Long Island City, New York
  - Lucas Research Inc., Morehead City, North Carolina
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University Diabetes & Endocrine Consultants, Chattanooga, Tennessee
  - Texas Diabetes & Endocrinology, PA, Austin, Texas
  - North Texas Endocrine Center, Dallas, Texas
  - Southern Endocrinology Associates, Mesquite, Texas
  - Diabetes & Glandular Disease Clinic, San Antonio, Texas
  - Diabetes & Endocrine Treatment Specialists, Sandy City, Utah
- Canada (7):
  - Centricity Research Calgary Endocrinology, Calgary, Alberta
  - BC Diabetes, Vancouver, British Columbia
  - Centricity Research Barrie Endocrinology, Barrie, Ontario
  - Centricity Research Vaughan Endocrinology, Concord, Ontario
  - Centricity Research Etobicoke Endocrinology, Etobicoke, Ontario
  - Centricity Research Toronto, Toronto, Ontario
  - Mount Sinai Hospital: Leadership Sinai Centre for Diabetes, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided